CLINICAL TRIAL: NCT02802618
Title: Interactive 3D Visualization Technique Used in Pulmonary Rehabilitation Programme in Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Interactive 3D Visualization Technique Used in Pulmonary Rehabilitation Programme in COPD
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska University Hospital (Other)
Collaborators: The Swedish Heart and Lung Association (Other); Landstingens Ömsesidiga Försäkringsbolag (Löf) (Unknown); Flemingsberg Science (Unknown); The Mats Kleberg Foundation (Unknown)
Responsible Party: Principal Investigator, Ulrika Einarsson, PhD, Karolinska University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2013/1276-31/3
Record Dates: First submitted 2016-05-27; First posted 2016-06-16 (Estimated); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Validity; Reliability; Rehabilitation; Translation; Education
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Interactive 3D visualization technique (Experimental): The pulmonary rehabilitation consists of exercise training during 10 weeks and a theoretic part presented with 3D technique.
  Patients randomized into education by 3D technique.
  Interventions: Other: Interactive 3D visualization technique
- Conventional technique (No Intervention): The pulmonary rehabilitation consists of exercise training during 10 weeks and a theoretic part presented with conventional technique. Patients randomized into education by conventional technique.

INTERVENTIONS:
Other: Interactive 3D visualization technique — The pulmonary rehabilitation consists of exercise training during two times/week for 10 weeks and a theoretic part presented with 3D visualization technique.
  Arms: Interactive 3D visualization technique

SUMMARY:
A new education material with 3D technique was developed, by integrating 3D technology in an existing evidence-based pulmonary educational program, to enable an increased personalized education within a group setting. The investigators believe that this educational model will lead to increased adherence to treatment, and suggested lifestyle changes, which in turn improves patients' HRQL

The purpose of this study was therefore to develop a pulmonary educational program in interactive 3D visualization technology and to evaluate differences between education with 3D technique or conventional technique in patient with COPD.

Furthermore the LCQ will be translated and culturally adapted into Swedish and tested for validity and reliability.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) is one of the major health scourges. In 2002 COPD was the fifth leading cause of death and estimates show that COPD becomes in 2030 the third leading cause of death worldwide. The dominant cause of COPD is tobacco smoking. COPD now affects men and women almost equally. The most common symptoms of COPD are breathlessness, excessive sputum production, and a chronic cough which causes decrease in health related quality of life (HRQL). Dyspnea and movement limitations are also common symptoms in patients with COPD and this often leads to reduced levels of physical activity, physical capacity and HRQL. The Leicester Cough Questionnaire (LCQ) is a valid evaluation tool for HRQL in patients with chronic cough. Currently no specific cough questionnaire exists in Swedish.

Pulmonary rehabilitation including education and exercise training improves health. The Physiotherapy department has conducted rehabilitation programs for patients with COPD since 1995. The COPD-program has several times been updated according to existing evidence.

Education in anatomy, physiology, physical therapy and self-training is a big part of the physical therapist's workday. The education imparts complex knowledge. It is demanding to mediate this as education is expected to raise the patient's desire to understand, create opportunities to understand and leave a lasting impression. In effective learning repetition, own search for information, stimulation, emotional impact and experience are important factors. Information technology is developing rapidly and patient's use of this technology is increasing. It is therefore essential that education is adapted to new requirements. Interactive 3 dimensional (3D) visualization techniques can be used to represent the human body. Interactive 3D technique used in patient education has not yet been studied.

A new education material with 3D technique was developed, by integrating 3D technology in an existing evidence-based pulmonary educational program, to enable an increased personalized education within a group setting. The investigators believe that this educational model will lead to increased adherence to treatment, and suggested lifestyle changes, which in turn improves patients' HRQL

In the current study it will be investigated whether och not there are differences between pulmonary educational program in interactive 3D visualization technology and in conventional technique in patients with COPD.

Furthermore the LCQ will be translated and culturally adapted into Swedish and tested for validity and reliability.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of chronic obstructive pulmonary disease (COPD)
* Stadium II-IV of COPD
* Must be able to comprehend the Swedish language

Exclusion Criteria:

* Not diagnosed with COPD
* Does not understand written and verbal Swedish

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2013-10; Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Improved health related quality of life | Change from Baseline health related quality of life at 10 weeks
  COPD Assessment Test

SECONDARY OUTCOMES:
Improved health related quality of life | Change from Baseline health related quality of life at 10 weeks
  S:t George´s Respiratory Questionnaire
Improved health related quality of life | Change from Baseline health related quality of life at 2 and 10 weeks
  Leicester Cough Questionnaire
Improved exercise self efficacy | Change from Baseline exercise self efficacy at 10 weeks
  SCI Exercise Self Efficacy Scale (SCI=Spinal Cord Injury)
Improved physical performance | Change from Baseline physical performance at 10 weeks
  JAMAR Hydraulic Hand Dynamometer
Improved physical performance | Change from Baseline physical performance at 10 weeks
  6 minute walk test
Attendance to rehabilitation programme | 10 weeks
  Attendance record
Improved knowledge of content in rehabilitation programme | Change from Baseline knowledge of content in rehabilitation programme at 6 months
  Questionaire
Compliance to treatment | 6 months
  Single question about compliance to treatment
Compliance to physical activity | 6 months
  Single question about compliance to physical activity
Visits to hospital, primary care | 6 months
  Single question about number of visits to hospital and primary care
Motivation with rehabilitation programme | 6 months
  Visual analog scale, focus group interview
Stimulation with the of rehabilitation programme | 6 months
  Visual analog scale, focus group interview

CONTACTS AND LOCATIONS:
Overall Officials: Ulrika Einarsson, PhD, Principal Investigator — Karolinska University Hospital
Locations (1):
- Department of physiotherapy, Karolinska University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Sonnerfors P, Nordlin AK, Nykvist M, Thunstrom U, Einarsson U. Interactive 3D visualisation technique used in pulmonary rehabilitation in chronic obstructive pulmonary disease: A randomised controlled study evaluating quality of life, compliance and use of health care. Digit Health. 2025 Jan 17;11:20552076241308940. doi: 10.1177/20552076241308940. eCollection 2025 Jan-Dec. PMID 39830146